CLINICAL TRIAL: NCT05712746
Title: Samtasu Post-marketing General Drug Use-results Survey in Patients with Volume Overload in Heart Failure.
Status: Recruiting | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 263-101-00017
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Samtasu for I.V. infusion — Drug: 8 mg/vial or 16mg/vial
  Dosage and Administration:
  The usual adult dosage of tolvaptan sodium phosphate is 16 mg once daily and intravenously infused over 1 hour.

SUMMARY:
To confirm the safety of tolvaptan sodium phosphate in patients with volume overload in heart failure.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* patients with a known hypersensitivity to Tolvaptan sodium phosphate or Tolvaptan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Japan with volume overload in heart failure who are planned to be newly started on Samtasu therapy
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety information (Adverse Event) | 14 days from the initiation of tolvaptan sodium phosphate treatment
  Any untoward medicinal occurrence in a patient or clinical study subject administered a Medicinal Product and which does not necessarily have a causal relationship with this treatment (see Annex Ⅳ, ICH-E2A Guideline).
  An Adverse Event can therefore be any unfavorable and unintended sign (e.g. abnormal laboratory finding), symptom, or disease temporally associated with the use of a Medicinal Product, whether or not it is considered causally related to the Medicinal Product.
Number of Special Situations | 14 days from the initiation of tolvaptan sodium phosphate treatment
  Collecting any Situations related to the use of an Otsuka product which may or may not be associated with an adverse event:
  * Maternal (pregnancy and breastfeeding) or paternal (via semen) exposure;
  * Exposure during breastfeeding;
  * Overdose/Incorrect dosage, misuse, abuse (e.g. patient sharing products);
  * Medication errors (e.g. patient took wrong dose);
  * Lack of therapeutic efficacy (e.g. the product doesn't work);
  * Occupational exposure (e.g.: nurse administering the product is exposed);
  * Cases of suspected transmission of infectious agents;
  * Use of suspected or confirmed falsified product(s) or quality defect of the product(s);
  * Withdrawal reactions;
  * Accidental exposure (e.g.: child takes parent's product);
  * Drug-drug/drug-food interactions;
  * Unintentional use of product in a non-approved population (e.g.: pediatric or geriatric population);
  * Disease progression/exacerbation of existing disease
Number of off-Label Use | 14 days from the initiation of tolvaptan sodium phosphate treatment
  Collecting any type of off-Label Use that refers to situations where a product is intentionally used for a medical purpose not in accordance with the authorized product information. Off-label use also includes the intentional use in nonauthorized population categories not indicated in the label.
Incidence of Serious Adverse Event (e.g. resulting in death or life-threatening) | 14 days from the initiation of tolvaptan sodium phosphate treatment
  Collecting the number of any adverse drug experience/event occurring at any dose which
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or prolonged of existing hospitalization
  * results in persistent or significant disability or incapacity
  * is a congenital anomaly/birth defect
  * is medically significant.
Incidence of Non-serious Adverse Events (i.e. all Adverse Events that do not meet the definition of a serious Adverse Event) | 14 days from the initiation of tolvaptan sodium phosphate treatment
  Collecting the number of non-serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Fukuta, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Pharmacovigilance Department, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No